CLINICAL TRIAL: NCT00489125
Title: Breast Clinic Strength and Range of Motion Study
Brief Title: Strength and Range of Motion in Women Undergoing Surgery for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CCCWFU 97305; P30CA012197 (NIH); CCCWFU-97305; CCCWFU-BG05-106
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: long-term effects secondary to cancer therapy in adults; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: physiologic testing — physical testing of range of motion, grip strength etc.

SUMMARY:
RATIONALE: Gathering information about strength and range of motion over time from women undergoing surgery for breast cancer may help doctors learn more about recovery from surgery and on-going care.

PURPOSE: This clinical trial is collecting information about strength and range of motion over time from women undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Collect data regarding diagnosis, type of surgery, receipt of adjuvant therapy, age, height, weight, waist circumference, arm strength, grip strength, shoulder range of motion, and physical activity participation from women undergoing surgery for breast cancer.
* Examine changes in physical activity participation, measures of body composition, shoulder range of motion, grip strength, and arm strength over time in these patients.
* Determine differences in changes in physical activity and indices of fitness according to type of surgery and adjuvant therapy.
* Examine relationships between exercise participation, fitness, and body composition over time.
* Correlate data with an ongoing randomized exercise trial that includes strength and flexibility assessments with no pre-surgery measures.

OUTLINE: This is a prospective, cohort study.

Patients submit data comprising demographic/medical information, anthropometrics (weight, height, waist circumference), grip strength, bicep strength, shoulder range of motion, and physical activity participation prior to surgery, at each surgical follow-up visit, and at 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer

  * Stage I-IV disease
* Planning to undergo surgery at the Comprehensive Cancer Center Breast Clinic at Wake Forest University Baptist Medical Center

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any woman treated in the Breast Clinic of WFUBMC with a diagnosis of stage 0-IV breast cancer and identified as a candidate by their surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2004-10-15 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Collection of data before surgery, at each follow-up visit, and at 2 years after surgery | approximately 2 years
Changes in physical activity participation, measures of body composition, shoulder range of motion, grip strength, and arm strength over time | approximately 2 years
Differences in changes in physical activity and indices of fitness according to type of surgery and adjuvant therapy | approximately 2 years
Relationships between exercise participation, fitness, and body composition over time | approximately 2 years
Correlation of data with an ongoing randomized exercise trial that includes strength and flexibility assessments with no pre-surgery measures | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Mihalko, PhD, Principal Investigator — Wake Forest University Health Sciences; Edward A. Levine, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States